CLINICAL TRIAL: NCT02775968
Title: Population Pharmacokinetics of Cephalosporins and Macrolides in Children With Community Acquired Pneumonia
Brief Title: Population Pharmacokinetics of Cephalosporins and Macrolides in Chinese Children With Community Acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Kunling Shen, Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: BCH_PPK001
Record Dates: First submitted 2016-05-11; First posted 2016-05-18 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Cephalosporins; Macrolides; Azithromycin; Erythromycin; Cefamandole; Moxalactam; Ceftriaxone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cephalosporins and Macrolide Antibiotics — The intervention drugs are prescribed by treating caregiver.
  Other Names: azithromycin; erythromycin; cefamandole; latamoxef; ceftriaxone

SUMMARY:
This study is based on the hypothesis that the pharmacokinetics of antibiotics in children is different from adults. Cephalosporins and macrolide antibiotics are the common drugs for children with community acquired pneumonia, the investigators aim to study the population pharmacokinetics of cephalosporins and macrolide antibiotics in children receiving the drug for treatment of community acquired pneumonia, and to correlate it with treatment effectiveness and incidence of adverse effects.

Potential Impact: This novel knowledge will allow better and more rational approaches to the treatment of community acquired pneumonia. It will also set the foundation for further studies that will be able to test improved therapies that may increase treatment response in vulnerable children.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-18 years old of both sexes, with a diagnosis of community acquired pneumonia and eligible for treatment with cephalosporins and macrolide antibiotics, as per current treatment protocols.
* Community acquired pneumonia diagnostic criteria: meet any one of the 1-4 following items plus the fifth item:

  * 1. With cough, expectoration, or pre-existing respiratory disease getting worse, and with purulent sputum with or without chest pain;
  * 2. Fever;
  * 3. With pulmonary consolidation and crackles;
  * 4. White blood cells>10×10^9/L or <4×10^9/L;
  * 5. X-ray on chest shows flake, patchy infiltrate shadows or interstitial changes, with or without pleural effusion.
* Informed consent signed by the parents, and consent or assent of the patients (according to age and consenting capacity).

Exclusion Criteria:

* It is unable to provide complete medical records or the current condition can not accept the diagnosis process.
* It does not agree to participate in this study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (1-18 years of age) receiving drugs per standard of care as prescribed by treating caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
maximum concentration (Cmax) | up to 4 weeks

SECONDARY OUTCOMES:
time to achieve maximum concentration (Tmax) | up to 4 weeks
absorption rate constant (ka) | up to 4 weeks
elimination rate constant (kel) | up to 4 weeks
half-life (t1/2) | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A-Dong Shen, Master, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China; Bao-Ping Xu, MD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China; China National Clinical Research Center for Respiratory Diseases
Locations (1):
- Beijing Children's Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jacqz-Aigrain E, Leroux S, Zhao W, van den Anker JN, Sharland M. How to use vancomycin optimally in neonates: remaining questions. Expert Rev Clin Pharmacol. 2015;8(5):635-48. doi: 10.1586/17512433.2015.1060124. Epub 2015 Aug 4. PMID 26289222
- [Background] Ho PL, Lo PY, Chow KH, Lau EH, Lai EL, Cheng VC, Kao RY. Vancomycin MIC creep in MRSA isolates from 1997 to 2008 in a healthcare region in Hong Kong. J Infect. 2010 Feb;60(2):140-5. doi: 10.1016/j.jinf.2009.11.011. Epub 2009 Dec 2. PMID 19961873
- [Background] Kearns GL, Abdel-Rahman SM, Alander SW, Blowey DL, Leeder JS, Kauffman RE. Developmental pharmacology--drug disposition, action, and therapy in infants and children. N Engl J Med. 2003 Sep 18;349(12):1157-67. doi: 10.1056/NEJMra035092. No abstract available. PMID 13679531